CLINICAL TRIAL: NCT04808115
Title: A Phase I Trial of Incorporating Natural Killer (K-NK) Cells for Patients With Chronic Myeloid Leukemia (CML) and Molecular Residual Disease After Tyrosine Kinase Inhibitor (TKI) Therapy
Brief Title: IIT PH1 KDS-1001 in Patients With CML
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant.
Sponsor: Duke University (Other)
Collaborators: Kiadis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106898
Record Dates: First submitted 2021-02-24; First posted 2021-03-22 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: CML (Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KDS-1001 (Experimental): KDS-1001 is infused on Day 1 of each 14 day cycle. Patients will receive 6 cycles of KDS-1001 treatment.
  Interventions: Drug: KDS-1001

INTERVENTIONS:
Drug: KDS-1001 — Cycles 1-6 (14 days per cycle)
  1 x 109/KDS-1001 cells/infusion administered on day 1 of each cycle

SUMMARY:
This open label, non-randomized, prospective phase I study is designed to evaluate if the addition of natural killer cell therapy (KDS-1001) to tyrosine kinase inhibitors (TKIs) for chronic myeloid leukemia (CML) patients with persistent or recurrent molecular residual disease (MRD) after at least one year of TKI therapy will allow patients to achieve RT-PCR negativity (MRD negative). This may have implications for future TKI cessation studies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-blast phase CML by standard definition. This should be confirmed by presence of the Philadelphia chromosome or variants of the (9;22) translocation by cytogenetics, FISH or with a positive RT-PCR for BCR-ABL. Repeat marrow not required for enrollment although documentation of current chronic phase disease is required.

   Chronic Phase CML is defined as follows:
   1. <15% blasts in peripheral blood and marrow
   2. <30% blasts plus promyelocytes in peripheral blood and marrow
   3. <20% basophils in peripheral blood
   4. >100 x 109/L platelets
   5. No evidence of extramedullary leukemic involvement with the exception of hepatosplenomegaly.

   Accelerated Phase CML is defined as follows:
   1. <30% blasts in blood, marrow or both
   2. No evidence of extramedullary leukemic involvement with the exception of hepatosplenomegaly.
2. > 18 years of age and able to provide informed consent
3. Patients must have been on TKI therapy for CML for at least 1 year prior to enrollment at minimum goal doses.

   Imatinib 300mg PO daily Dasatinib 70mg PO daily Nilotinib 200mg PO BID Bosutinib 300mg PO daily Ponatinib 30mg PO daily Lower than goal doses are allowed IF documented by the treating physician that the goal dose was not tolerable due to toxicity.
4. Patient must have been on their most recent TKI consistently for at least 6 months prior to enrollment on study
5. Must be expected to remain on current TKI for at least 6 months following last infusion, unless there is progression of disease.
6. Detectable BCR-ABL transcripts measured by RT-PCR at a CLIA-approved laboratory and reported on the IS with a value of >0.01% within 28 days prior to study enrollment. The chosen RT-PCR test must be sensitive enough to detect a 4.5 log reduction in BCR/ABL transcripts measured in peripheral blood.
7. Performance status must be ECOG PS 0, 1, or 2.
8. Woman of childbearing potential and is willing to use 2 highly effective methods of contraception while receiving study treatment and for an additional 3 months after the last dose of protocol-specified therapy. Male who has a female partner of childbearing potential, and is willing to use 2 highly effective forms of contraception for at least an additional 3 months after the last dose of protocol-specified therapy.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. Current blast crisis phase disease by standard definition from the NCCN
2. Pregnant or lactating females
3. On other investigational agents for CML within 4 weeks of study enrollment
4. Platelets of <50,000/mm3, ANC <500/mm3 or hemoglobin < 7.5 g.dL
5. Abnormal screening laboratory values as defined below:

   1. AST (SGOT) and/or ALT (SGPT) and/or alkaline phosphatase ≥ 5 x upper limit of normal (ULN)
   2. Total bilirubin >1.5 x ULN (unless related to Gilbert´s or Meulengracht disease or leukemic infiltration)
   3. Creatinine ≥ 3 ULN or creatinine clearance < 50 mL/min (calculated)
   4. Those with residual toxicity of >grade 1 from prior therapy in areas that may be expected to worsen over time; those with residual toxicities of grade 2 which are stable prior to enrollment and the natural history of which would be expected to be 'no change' over time are allowed; those with grade 3 or 4 residual toxicities are not.
6. Positive test for human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS)
7. Positive hepatitis B virus (HBV) or hepatitis C virus (HCV) indicating acute or chronic infection (those with prior infection that is now post treatment and PCR negative are allowed)
8. Current use of immunosuppressive medications at the time of study enrollment and within 2 weeks of any study treatments, except:

   1. Intranasal, inhaled, topical steroids, or local steroid injection
   2. Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or equivalent
   3. Steroids as premedication for hypersensitivity reactions at physiologic doses ≤10 mg/day of prednisone or equivalent
9. Patients with other major medical or psychiatric illnesses, which the treating physician feels, could seriously compromise tolerance or compliance to this protocol.
10. Diagnosis of prior immunodeficiency or organ transplant requiring immunosuppressive therapy
11. Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, deep vein thrombosis, or symptomatic pulmonary embolism
12. Known prior or suspected hypersensitivity to study drugs or any component in their formulations
13. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
14. Diagnosis of any other malignancy within 3 years, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the breast or of the cervix, low grade prostate cancer on surveillance without any plans for treatment intervention, or prostate cancer that has been adequately treated with prostatectomy or radiotherapy and currently with no evidence of disease or symptoms
15. Active infection requiring systemic therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Molecular Response | End of Treatment up to two weeks
  At least one (1) log reduction in IS OR negative to at least MR4.5 via PCR-based testing
Safety of KDS-1001 | End of Study up to two years
  Number of adverse events as measured by self report

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Rein, MD, Principal Investigator — Assistant Professor of Medicine, Hematologic Malignancies & Cell Therapy

IPD SHARING:
Plan to Share IPD: No